CLINICAL TRIAL: NCT07077759
Title: An Online Self-compassion Intervention for Anxiety and Depression in Fathers of Infants: A Feasibility Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Principal Investigator, Dr Polly MA Haixia, Assistant Professor, Hong Kong Metropolitan University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HE-RD/2025/1.8
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Postpartum Depression (PPD)
Keywords: Paternal perinatal depression; father; self-compassion
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: non-RCT with a waiting-list control group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online self-compassion intervention (Experimental): Participants in the self-compassion group will receive five consecutive weekly sessions intervention.
  Interventions: Other: Online self-compassion intervention
- Control group (No Intervention): Participants in the waiting-list control group will receive the same training after the completion of the intervention at a 2-month follow-up.

INTERVENTIONS:
Other: Online self-compassion intervention — Participants in the intervention group will receive five consecutive weekly sessions, with each session lasting 2 hours (totaling 10 hours). Each session will include an introduction, guided exercises, group discussions and home practice.
  Arms: Online self-compassion intervention

SUMMARY:
To investigate the feasibility, acceptability, and preliminary effectiveness of an online mindfulness and self-compassion intervention for the mental health in fathers experiencing paternal perinatal depression (PPD).

DETAILED DESCRIPTION:
The pilot non-RCT will be assessed using an online survey and semi-structured individual interviews. Preliminary effectiveness measures include self-compassion, emotion regulation, resilience, parenting sense of competence, parental stress, marital satisfaction, insomnia, generalized anxiety, and PPD measured at baseline, immediate post-intervention, and 2-month follow-up. Mixed-effects models will test changes between groups, while directed content analysis will be employed for qualitative data.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or above
* the biological father who is expecting or the biological father of infants within 24 months old
* experienced mild to moderate anxiety (5 ≤ GAD ≤14) or depression symptoms (5≤ PHQ ≤ 19)
* sufficient comprehension of Cantonese
* currently live in Hong Kong
* able to provide informed consent

Exclusion Criteria:

* currently experiencing psychosis
* having an intellectual disability
* experiencing current suicidal ideation
* participation in a similar study or received similar services in the past year

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Paternal perinatal depression | From enrollment to the end of treatment at 2 months.
  Paternal perinatal depression will be measured using the Chinese version of the 9-item Patient Health Questionnaire (PHQ-9). Items are rated on a 4-point Likert scale ranging from 0 (not at all) to 3 (nearly every day). The total score ranges from 0 to 27, with higher total scores indicating higher levels of depressive symptoms. The scale is reliable in the Chinese population (Cronbach's α = 0.82).
Anxiety | From enrollment to the end of treatment at 2 months.
  Anxiety symptoms will be measured using the 7-item Generalized Anxiety Disorder-7 (GAD-7). Items are rated on a 4-point Likert scale ranging from 0 (not at all) to 3 (nearly every day). The total score ranges from 0 to 21, with higher total scores indicating higher levels of anxiety symptoms.

SECONDARY OUTCOMES:
Emotion regulation | From enrollment to the end of treatment at 2 months
  Emotion regulation will be measured by the 10-item Emotion Regulation Questionnaire (ERQ). It includes two subscales: Cognitive reappraisal and expressive suppression. Items are rated on a 7-point scale (1=Strongly Disagree to 7=Strongly Agree). The total score for cognitive reappraisal ranges from 0 to 42, and the total score for expressive supression ranged from 0 to 28. Higher scores mean more frequent use of that strategy.The Cronbach's alpha was 0.82 and 0.77 for cognitive reappraisal and suppression, respectively.
Self-compassion | From enrollment to the end of intervention at 2 months
  Self-compassion will be measured using the 12-item short version of the self-compassion scale (SCS). Items are rated on a 5-point Likert scale ranging from 1 (Almost Never) to 5 (Almost Always). The total score ranged from 12 to 60, with higher score indicating higher level of self-compassion. The scale has demonstrated good internal consistency in Chinese sexual minorities (Cronbach's alpha = 0.87)
Resilience | From enrollment to the end of treatment at 2 months.
  Resilience will be measured by the six-item brief resilience scale (BRS). Items are rated on a five-point Likert scale ranging from 1 (Strongly Disagree) to 5 (Strongly Agree). The total score ranges from 6 to 30, with higher score indicating higher level of resilience.
insomnia | From enrollment to the end of treatment at 2 months.
  Insomnia will be measured using the 7-item Insomnia Severity Index (ISI). Items are measured on five point likert scale (0-4). The total score of 0-28, with higher scores meaning worse insomnia.
Parent sense of competency | From enrollment to the end of treatment at 2 months.
  Participant's sense of parent competency will be measured using the 17-item Parent Sense of Competency Scale (PSOC). Items are rated on a 6 point Likert scale anchored by 1 = "Strongly Disagree" and 6 = "Strongly Agree". The total score ranged from 17 to 102, with higher score indicating high level of parent competency.
Parental stress | From enrollment to the end of treatment at 2 months.
  Parental stress will be measured using the 17-item of the Chinese version of Parental Stress Scale (PSS). Items are raged on a 6-point Likert scale (1 = strongly disagree, 6 = strongly agree). The total score ranges from 17 to 102, with higher score indicating higher level of parental stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Metropolitan University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No